CLINICAL TRIAL: NCT00835185
Title: Open Label, Multicenter, Phase II Study Evaluating the Efficacy and Safety of IMC-11F8 in Combination With 5-FU/FA and Oxaliplatin (mFOLFOX-6) in Patients With Treatment-naïve, Locally-advanced or Metastatic Colorectal Cancer
Brief Title: Study of IMC-11F8 in Participants With Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13926; 2006-003147-23 (EudraCT Number); CP11-0602 (Other: ImClone Systems); I4X-IE-JFCD (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Antibodies, Monoclonal; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — necitumumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-11F8 (necitumumab) /mFOLFOX-6 regimen (Experimental): Participants will receive IMC-11F8 (necitumumab) once every 2 weeks in combination with the mFOLFOX-6 regimen (oxaliplatin/5-FU/FA)
  Interventions: Biological: IMC-11F8 (necitumumab); Drug: Oxaliplatin; Drug: Folinic acid (FA); Drug: 5-FU

INTERVENTIONS:
Biological: IMC-11F8 (necitumumab) — IMC-11F8 800 milligrams (mg) intravenous (IV) infusion over 50 minutes on Day 1
  Other Names: Necitumumab; IMC-11F8; LY3012211; Portrazza®
Drug: Oxaliplatin — Oxaliplatin 85 milligrams per meter square (mg/m²) IV infusion over 2 hours on Day 1
Drug: Folinic acid (FA) — FA 400 mg/m² IV infusion bolus injection
Drug: 5-FU — 5-FU 400 mg/m² as a bolus followed by 2400 mg/m² IV continuous infusion over 46 hours

SUMMARY:
The purpose of this study is to determine if IMC-11F8 in combination with chemotherapy is effective in treating colorectal cancer (CRC).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the anti-tumor activity (best overall response) of the anti-epidermal growth factor receptor (EGFR) monoclonal antibody IMC-11F8 administered in combination with mFOLFOX-6 chemotherapy regimen in treatment-naive, locally-advanced or metastatic CRC participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, EGFR-detectable or EGFR-undetectable CRC
* Locally-advanced unresectable or metastatic adenocarcinoma of the colon or rectum
* At least 1 unidimensional-measurable target lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI); target lesion(s) must not lie within an irradiated area
* Age ≥18 years
* Life expectancy of ≥6 months
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 at study entry
* Adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥1.5 x 10^9 liter (L), hemoglobin ≥10 grams per deciliter (g/dL), and platelets ≥100 x 10^9/L
* Adequate hepatic function as defined by a total bilirubin ≤1.5 milligrams per deciliter (mg/dL), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN) (or 5.0 x ULN in the case of liver metastases), and alkaline phosphatase (AP) ≤2.5 x ULN (or 5.0 x ULN in the case of liver metastases)
* Adequate renal function as defined by a serum creatinine ≤1.5 x ULN, creatinine clearance ≥ 60 milliliters per minute (mL/min), or serum albumin ≥lower limit of normal (LLN)
* Participant's relevant toxicities/effects of prior therapy [surgery/radiation therapy (RT)] must have recovered to a stable or chronic level
* Participant agrees to use adequate contraception during the study period and for 4 weeks after the last dose of study treatment. Participants must notify the principal investigator if they themselves or their partner becomes pregnant.
* Participant has provided signed Informed Consent

Exclusion Criteria:

* Has received prior systemic chemotherapy for locally-advanced unresectable or metastatic CRC.
* Has received prior radiotherapy to >25% of bone marrow
* Has documented and/or symptomatic brain metastases
* Has participated in clinical studies of non-approved experimental agents or procedures within 12 weeks of study entry
* Has received previous therapy with monoclonal antibodies
* Has received previous therapy with any agent that targets the EGFR
* Has serious concomitant medical conditions including active uncontrolled infection or cardiac disease, which in the opinion of the investigator, could compromise the participant or study.
* On chronic non-topical corticosteroid treatment for >6 months at doses >10 milligrams per day (mg/day) of prednisolone or equivalent before study entry, which in the opinion of the investigator could compromise the participant or the study
* Has a known dihydropyrimidine dehydrogenase deficiency
* Has a known allergy to any of the treatment components
* Has an acute or subacute intestinal occlusion
* Has peripheral neuropathy ≥Grade 2
* Has a history of other malignancies, with the exception of curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix
* If female, is pregnant (confirmed by urine or serum beta human chorionic gonadotropin test) or breast-feeding
* Has received a prior autologous or allogeneic organ or tissue transplantation
* Has interstitial pneumonia or interstitial fibrosis of the lung
* Has pleural effusion or ascites that causes ≥Grade 2 dyspnea
* Has psychological, familial, sociological, or geographical conditions which do not permit adequate study follow-up, compliance with the protocol, or signature of Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-08; Primary Completion 2010-01 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- Belgium (2):
  - ImClone Investigational Site, Brussels
  - ImClone Investigational Site, Haine-Saint-Paul
- Spain (3):
  - ImClone Investigational Site, Barcelona
  - ImClone Investigational Site, Madrid
  - ImClone Investigational Site, Valencia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with known best overall response and off study treatment were considered to be completed.
Groups:
- IMC-11F8 (Necitumumab) + mFOLFOX-6: On Day 1 of each 2-week cycle, each participant received IMC-11F8 (necitumumab) in combination with the mFOLFOX-6 regimen (oxaliplatin/5-FU/FA) in the order shown:
  * 800 milligrams (mg) IMC-11F8 intravenous (IV) infusion over 50 minutes
  * 85 milligrams per meter square (mg/m²) oxaliplatin IV infusion over 2 hours
  * 400 mg/m² folinic acid
  * 400 mg/m² 5-FU as an IV bolus injection; and immediately followed by
  * A 46-hour continuous IV infusion of 5-FU at 2400 mg/m² All treatments were administered every 2 weeks until disease progression, the development of unacceptable toxicity, noncompliance, withdrawal of consent or until other criteria for treatment discontinuation were met.
Period: Overall Study
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Started | 44
Received at Least 1 Dose of Study Drug | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received any quantity of study drug.
Groups:
- IMC-11F8 (Necitumumab) + mFOLFOX-6: On Day 1 of each 2-week cycle, each participant received IMC-11F8 (necitumumab) in combination with the mFOLFOX-6 regimen (oxaliplatin/5-FU/FA) in the order shown:
  * 800 mg IMC-11F8 IV infusion over 50 minutes
  * 85 mg/m² oxaliplatin IV infusion over 2 hours
  * 400 mg/m² folinic acid
  * 400 mg/m² 5-FU as an IV bolus injection; and immediately followed by
  * A 46-hour continuous IV infusion of 5-FU at 2400 mg/m² All treatments were administered every 2 weeks until disease progression, the development of unacceptable toxicity, noncompliance, withdrawal of consent, investigator decision, or until other criteria for treatment discontinuation were met.
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 13
  Spain | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response )
Description: CR and PR defined using Response Evaluation Criteria In Solid Tumors (RECIST) version (v) 1.0 criteria. CR was defined as the disappearance of all target and non-target lesions and PR defined as a ≥30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD. Percentage of participants was calculated as: (total number of participants with CR or PR from start of the treatment until disease progression or recurrence) / (total number of participants treated) * 100.
Time Frame: Up to 30 Months
Population: All enrolled participants who received any quantity of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 44
percentage of participants | 63.6 [47.8 to 77.6]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from the date of first dose to the date of death from any cause. OS was estimated by the Kaplan-Meier method. Participants who were alive at the time of the data inclusion cutoff or lost to follow-up, OS was censored at the last contact.
Time Frame: First dose to date of death from any cause up to 30 months
Population: All enrolled participants who received any quantity of study drug. Participants censored =14.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 44
months | 22.5 [11.0 to 30.0]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from date of first dose to the first observation of disease progression or death due to any cause. Progressive disease (PD) was determined using RECIST v1.0 criteria. PD was defined as ≥20% increase in the sum of LD of target lesions, taking as reference the smallest sum of the LD recorded since treatment started or the appearance of new lesions and/or unequivocal progression of existing nontarget lesions. PFS was estimated by the Kaplan-Meier method. Participants who had no PD or death at the time of the data inclusion cutoff, PFS was censored at their last tumor assessment prior to the earliest of the following events: 2 or more missed visits, additional cancer treatment or the end of the follow-up period.
Time Frame: First dose to measured PD or death up to 30 months
Population: All enrolled participants who received any quantity of study drug. Participants censored =13.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 44
months | 10.0 [7.0 to 12.0]

4. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs) or Death
Description: The number of participants who experienced AEs, SAEs or death during the study and within 30 days of last dose. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: First dose to end of treatment and 30-day post treatment follow-up up to 31 months
Population: All enrolled participants who received any quantity of study drug.
Measure: Number; unit: participants
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 44
participants
  AEs | 44
  SAEs | 16
  Deaths | 3

5. Secondary Outcome: Duration of Response
Description: The duration of response was defined as the time from first confirmed CR or PR to the first time of PD or death due to any cause. CR, PR and PD were defined using RECIST v1.0 criteria. CR was defined as the disappearance of all target and non-target lesions; PR was defined as a ≥30% decrease in the sum of the LD of the target lesions, taking as reference the baseline sum of the LD; PD was defined as a ≥20% increase in the sum of LD of target lesions, taking as reference the smallest sum of the LD recorded since treatment started or the appearance of new lesions and/or unequivocal progression of existing nontarget lesions. Participants with CR or PR who had no PD or death at the time of the data inclusion cutoff, the duration of response was censored at their last contact.
Time Frame: Time of response to time of measured PD or death up to 30 months
Population: All enrolled participants who received any quantity of study drug and had confirmed CR or PR. Participants censored =2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 28
months | 10.0 [7.0 to 16.0]

6. Secondary Outcome: Serum Anti-IMC-11F8 Antibody Assessment (Immunogenicity)
Description: A participant was considered to have an anti-IMC-11F8 response if there were 2 consecutive positive samples or if the final sample tested is positive. Participants with a baseline sample positive for anti-IMC-11F8 antibodies were considered unevaluable for immunogenicity. A sample was considered positive for IMC-11F8 antibodies if it exhibited a post-baseline treatment emergent antibody level that exceeded the upper 95% confidence interval of the mean determined from the normal anti-IMC 11F8 level found in healthy treatment-naïve individuals.
Time Frame: Baseline up to last day of treatment plus 45 days after last treatment (127 weeks)
Population: All participants who received any amount of study drug and were IMC-11F8 antibody negative at baseline.
Measure: Number; unit: participants
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 42
participants | 4

7. Secondary Outcome: Maximum Concentration (Cmax) of IMC-11F8 at Study Day 1 of Cycle 1
Time Frame: Cycle 1 Day 1 predose, immediately after infusion, and 1, 2, 4, 24, 72, 96, 144, 168 and 236 hours postdose
Population: All enrolled participants who received any quantity of study drug and had pharmacokinetic (PK) data available to calculate Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Groups:
- IMC-11F8 (Necitumumab) + mFOLFOX-6: On Day 1 of Cycle 1, each participant received IMC-11F8 (necitumumab) in combination with the mFOLFOX-6 regimen (oxaliplatin/5-FU/FA) in the order shown:
  * 800 mg IMC-11F8 IV infusion over 50 minutes;
  * 85 mg/m² oxaliplatin IV infusion over 2 hours;
  * 400 mg/m² folinic acid;
  * 400 mg/m² 5-FU as an IV bolus injection; and immediately followed by
  * A 46-hour continuous IV infusion of 5-FU at 2400 mg/m². All treatments were administered every 2 weeks until disease progression, the development of unacceptable toxicity, noncompliance, withdrawal of consent, investigator decision or until other criteria for treatment discontinuation were met.
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 39
micrograms/milliliter (µg/mL) | 344 (46)

8. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity [AUC(0-∞)] of IMC-11F8 at Study Day 1 of Cycle 1
Time Frame: Cycle 1 Day 1 predose, immediately after infusion, and 1, 2, 4, 24, 72, 96, 144, 168 and 236 hours postdose
Population: All enrolled participants who received any quantity of study drug and had PK data available to calculate AUC(0-∞).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter (µg*h/mL)]
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 17
micrograms*hour/milliliter (µg*h/mL)] | 39400 (35)

9. Secondary Outcome: Half-Life (t1/2) of IMC-11F8 at Study Day 1 of Cycle 1
Description: The t1/2 is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: Cycle 1 Day 1 predose, immediately after infusion, and 1, 2, 4, 24, 72, 96, 144, 168 and 236 hours postdose
Population: All enrolled participants who received any quantity of study drug and had PK data available to calculate t1/2.
Measure: Geometric Mean (Full Range); unit: hours (h)
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 17
hours (h) | 142 [99.8 to 299]

10. Secondary Outcome: Clearance (CL) of IMC-11F8 at Study Day 1 of Cycle 1
Description: CL is the volume of plasma (or blood) from which the drug is completely removed, or cleared, in a given time.
Time Frame: Cycle 1 Day 1 predose, immediately after infusion, and 1, 2, 4, 24, 72, 96, 144, 168 and 236 hours postdose
Population: All enrolled participants who received any quantity of study drug and had PK data available to calculate CL.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters/hour (mL/h)
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 17
milliliters/hour (mL/h) | 20.3 (35)

11. Secondary Outcome: Volume of Distribution (Vss) of IMC-11F8 at Study Day 1 of Cycle 1
Description: Vss is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug at steady-state.
Time Frame: Cycle 1 Day 1 predose, immediately after infusion, and 1, 2, 4, 24, 72, 96, 144, 168 and 236 hours postdose
Population: All enrolled participants who received any quantity of study drug and had PK data available to calculate Vss.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters (mL)
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 17
milliliters (mL) | 3660 (32)

12. Secondary Outcome: Cmax at Study Day 1 of Cycles 2 Through 6
Time Frame: Day 1 Cycles 2 through 6 predose and 1 hour postdose
Population: Zero participants were analyzed, Cmax results were not collected.
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 0

13. Secondary Outcome: Area Under the Curve (AUC) at Study Day 1 of Cycles 2 Through 6
Time Frame: Day 1 Cycles 2 through 6 predose and 1 hour postdose
Population: Zero participants were analyzed, AUC results were not collected.
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 0

14. Secondary Outcome: t1/2 at Study Day 1 of Cycles 2 Through 6
Time Frame: Day 1 Cycles 2 through 6 predose and 1 hour post dose
Population: Zero participants were analyzed, t1/2 results were not collected.
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 0

15. Secondary Outcome: CL at Study Day 1 of Cycles 2 Through 6
Time Frame: Day 1 Cycles 2 through 6 predose and 1 hour postdose
Population: Zero participants were analyzed, CL results were not collected.
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 0

16. Secondary Outcome: Vss at Study Day 1 of Cycles 2 Through 6
Time Frame: Day 1 Cycles 2 through 6 predose and 1 hour postdose
Population: Zero participants were analyzed, Vss results were not collected.
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 0

17. Secondary Outcome: Change From Baseline in Tumor Size
Time Frame: Baseline, 29 Months
Population: Zero participants were analyzed, the outcome measure was registered in error.
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 0

18. Secondary Outcome: Kirsten Rat Sarcoma (KRAS) Mutation Status
Description: Tumor tissues collected prior to study drug administration were evaluated for the presence or absence of KRAS mutations by a retrospective analysis.
Time Frame: Baseline
Population: All enrolled participants who had assessment of tumor tissue samples at baseline.
Measure: Number; unit: participants
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Number analyzed (Participants) | 25
participants
  KRAS Mutation Positive | 9
  KRAS Mutation Negative | 16

ADVERSE EVENTS:
Groups:
- IMC-11F8 (Necitumumab) + mFOLFOX-6: On Day 1 of each 2-week cycle, each participant received IMC-11F8 (necitumumab) in combination with the mFOLFOX-6 regimen (oxaliplatin/5-FU/FA) in the order shown:
  * 800 mg IMC-11F8 IV infusion over 50 minutes;
  * 85 mg/m² oxaliplatin IV infusion over 2 hours;
  * 400 mg/m² folinic acid;
  * 400 mg/m² 5-FU as an IV bolus injection; and immediately followed by
  * A 46-hour continuous IV infusion of 5-FU at 2400 mg/m². All treatments were administered every 2 weeks until disease progression, the development of unacceptable toxicity, noncompliance, withdrawal of consent, investigator decision, or until other criteria for treatment discontinuation were met.
Arm/Group | IMC-11F8 (Necitumumab) + mFOLFOX-6
Serious Adverse Events (participants affected / at risk) | 16/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-11F8 (Necitumumab) + mFOLFOX-6 (N=44)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (5)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Medical device complication (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-11F8 (Necitumumab) + mFOLFOX-6 (N=44)
Anaemia (Blood and lymphatic system disorders) | 9 (15)
Neutropenia (Blood and lymphatic system disorders) | 23 (61)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (30)
Conjunctivitis (Eye disorders) | 11 (17)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 13 (18)
Diarrhoea (Gastrointestinal disorders) | 24 (60)
Dyspepsia (Gastrointestinal disorders) | 5 (9)
Nausea (Gastrointestinal disorders) | 17 (33)
Oesophagitis (Gastrointestinal disorders) | 3 (4)
Rectal tenesmus (Gastrointestinal disorders) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 8 (16)
Vomiting (Gastrointestinal disorders) | 16 (31)
Asthenia (General disorders) | 36 (110)
Fatigue (General disorders) | 4 (5)
Mucosal inflammation (General disorders) | 19 (67)
Pyrexia (General disorders) | 9 (15)
Hypersensitivity (Immune system disorders) | 3 (4)
Paronychia (Infections and infestations) | 16 (45)
Respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Weight decreased (Investigations) | 14 (20)
Weight increased (Investigations) | 7 (11)
Decreased appetite (Metabolism and nutrition disorders) | 18 (34)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5)
Dysaesthesia (Nervous system disorders) | 13 (46)
Dysgeusia (Nervous system disorders) | 7 (12)
Headache (Nervous system disorders) | 4 (5)
Neuropathy peripheral (Nervous system disorders) | 3 (5)
Neurotoxicity (Nervous system disorders) | 9 (15)
Paraesthesia (Nervous system disorders) | 16 (50)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (54)
Insomnia (Psychiatric disorders) | 3 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (11)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (10)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 (24)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 31 (104)
Skin fissures (Skin and subcutaneous tissue disorders) | 10 (23)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.